CLINICAL TRIAL: NCT04914000
Title: Motivating a Spectrum of Cancer Patients to Quit Smoking: Intervention Development and Feasibility
Brief Title: Motivating a Spectrum of Cancer Patients to Quit Smoking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MCC-19733; 1R03CA227044-01A1 (NIH)
Record Dates: First submitted 2019-04-12; First posted 2021-06-04 (Actual); Results first posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-02

CONDITIONS: Cancer; Smoking
MeSH Terms: conditions — Neoplasms; Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Self Help Materials (Experimental): Participants will receive a smoking cessation booklet/pamphlet corresponding to their cancer type.
  Interventions: Behavioral: Self-help Materials

INTERVENTIONS:
Behavioral: Self-help Materials — Self-help booklet targeted by cancer type to increase smoking cessation motivation

SUMMARY:
This study will assess feasibility and acceptability of an intervention designed to increase smoking cessation motivation among patients with a cancer not widely known to be smoking related.

ELIGIBILITY:
Inclusion Criteria:

* Smoking at least 1 cigarette in previous 30 days
* Diagnosis of breast, colorectal, gynecological, skin melanoma, or bladder cancer within the last 6 months
* Able to read/write English
* Able to give informed consent
* Not currently enrolled in a smoking cessation program

Exclusion Criteria:

* Having distant metastases
* Male patients with breast cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2022-04-13 (Actual); Study Completion 2022-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Martinez, Ph.D., Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Self Help Materials
Started | 53
Completed | 44
Not Completed | 9
Not completed — Lost to Follow-up | 8
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Self Help Materials
Number analyzed (Participants) | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 37
  >=65 years | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 51
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 53
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 53

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Consent to Participate in the Study- Feasibility
Description: Number of participants who consent to participate in the study
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Self Help Materials
Number analyzed (Participants) | 53
Participants | 53

2. Primary Outcome: Number of Participants That Complete 1-week Follow-up Assessments - Feasibility
Description: Number of participants who complete 1-week follow-up assessments
Time Frame: 1-week post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Self Help Materials
Number analyzed (Participants) | 48
Participants | 46

3. Primary Outcome: Number of Participants That Complete 1 Month Follow-up Assessments - Feasibility
Description: Number of participants who complete 1-month follow-up assessments
Time Frame: 1-month post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Self Help Materials
Number analyzed (Participants) | 48
Participants | 44

4. Primary Outcome: Number of Participants Who Read the Booklet - Demand - 1 Week Post Treatment
Description: Number of study participants who read the booklet
Time Frame: 1-week post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Self Help Materials
Number analyzed (Participants) | 46
Participants | 38

5. Primary Outcome: Number of Participants Who Read the Booklet - Demand - 1 Month Post Treatment
Description: Number of study participants who read the booklet
Time Frame: 1-month post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Self Help Materials
Number analyzed (Participants) | 44
Participants | 42

6. Primary Outcome: Acceptability
Description: Treatment satisfaction measured with 8 items adapted from the Client Satisfaction Questionnaire, values between 8 and 32, with higher scores mean a better outcome.
Time Frame: 1-month post-treatment
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Self Help Materials
Number analyzed (Participants) | 40
score on a scale | 24.43 [8 to 32]

7. Secondary Outcome: Motivation to Quit Smoking Assessed With the Contemplation Ladder
Description: Changes in motivation to quit smoking will be assessed using the Contemplation Ladder. This is a validated measure for the assessment of readiness to quit smoking on a scale from 0 to 10. Higher scores indicate greater motivation to quit smoking.
Time Frame: Baseline, 1-week post-treatment, 1-month post-treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Self Help Materials
Number analyzed (Participants) | 48
units on a scale
  Basline | 7.35 (2.22)
  1 week post treatment | 7.58 (2.58)
  1 month post treatment | 7.79 (2.41)

8. Secondary Outcome: Motivation to Quit Smoking Assessed With the Short Form of the Smoking Abstinence-related Motivational Engagement (ARME).
Description: Changes in motivation to quit smoking will be assessed using the short form of the smoking abstinence-related motivational engagement (ARME), which is a valid and reliable measure of cessation motivation that includes 5 items related to the smokers' daily experience with scores ranging from 5 to 35. Higher scores indicate greater motivation to quit smoking.
Time Frame: Baseline, 1-week post-treatment, 1-month post-treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Self Help Materials
Number analyzed (Participants) | 48
score on a scale
  Baseline | 23.41 (7.77)
  1 Week Post Treatment | 24.59 (8.05)
  1 Month Post Treatment | 24.11 (7.96)

9. Secondary Outcome: Participants Change in Motivation - Action Stage
Description: Changes in motivation to quit smoking will be assessed using the Stages of Change algorithm (SOC). This is a widely used measure for the assessment of readiness to quit smoking.
Time Frame: Baseline, at 1 week and 1 month post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Self Help Materials
Number analyzed (Participants) | 47
Participants
  Baseline | 4
  1 week post treatment | 6
  1 month post treatment | 12

10. Secondary Outcome: Motivation to Quit Smoking Assessed With the Number of Visits to the Study Website
Description: A personal code will be able to track the number of participants who visited the study website where participants will find existing smoking cessation resources. This will be considered a behavioral indicator of motivation to quit smoking.
Time Frame: 1-month post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Self Help Materials
Number analyzed (Participants) | 48
Participants | 1

11. Secondary Outcome: Motivation to Quit Smoking Assessed by Contact With the Tobacco Treatment Specialist - 1 Week
Description: Participants will be asked if they have contacted the tobacco treatment specialist or if they would like us to make a referral for them. This will be considered a behavioral indicator of motivation to quit smoking.
Time Frame: At 1 Week Post Treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Self Help Materials
Number analyzed (Participants) | 46
Participants
  Contacted Smoking Cessation Program | 2
  Requested a Referral | 10

12. Secondary Outcome: Motivation to Quit Smoking Assessed by Contact With the Tobacco Treatment Specialist - 1 Month
Description: as for outcome 11
Time Frame: At 1 Month Post Treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Self Help Materials
Number analyzed (Participants) | 43
Participants
  Contacted Smoking Cessation Program | 3
  Requested a Referral | 10

13. Secondary Outcome: Participants That Had a Quit Attempt - 1 Week
Description: Number of participants that had a quit attempt that lasted at least 24 hours (at the 1-week assessment)
Time Frame: At 1 Week Post Treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Self Help Materials
Number analyzed (Participants) | 46
Participants | 15

14. Secondary Outcome: Participants That Had a Quit Attempt - 1 Month
Description: Number of participants that had a quit attempt that lasted at least 24 hours
Time Frame: At 1 Month Post Treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Self Help Materials
Number analyzed (Participants) | 44
Participants | 25

15. Secondary Outcome: Motivation to Quit Smoking Assessed With the Number of Quit Attempts - 1 Month
Description: Number of times participants quit smoking in the last 30 days (at the 1-month assessment).
Time Frame: At 1 Month Post Treatment
Measure: Mean (Standard Deviation); unit: Times participants quit smoking
Arm/Group | Self Help Materials
Number analyzed (Participants) | 44
Times participants quit smoking | 6.74 (10.70)

16. Secondary Outcome: Number of Participants Reporting 7-day Point Prevalence Abstinence
Description: Smoking abstinence will be determined by a self-report of not smoking in the last 7 days
Time Frame: 1-week post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Self Help Materials
Number analyzed (Participants) | 46
Participants | 6

17. Secondary Outcome: Number of Participants Reporting 30-day Point Prevalence Abstinence
Description: Smoking abstinence will be determined by a self-report of not smoking in the last 30 days
Time Frame: 1-month post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Self Help Materials
Number analyzed (Participants) | 44
Participants | 12

ADVERSE EVENTS:
Time Frame: Adverse Events were not collected
Description: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed
Arm/Group | Self Help Materials
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/00/NCT04914000/Prot_SAP_000.pdf
  • Informed Consent Form (2021-05-17): https://cdn.clinicaltrials.gov/large-docs/00/NCT04914000/ICF_001.pdf